CLINICAL TRIAL: NCT03501303
Title: A Nordic, Multicentre, Prospective, Randomized, Register Based, Clinical Trial on No-touch Vein Graft (NT-graft) in Coronary Surgery
Brief Title: A Clinical Trial on No-touch Vein Graft (NT-graft) in Coronary Surgery
Acronym: SWEDEGRAFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U-2015-477
Record Dates: First submitted 2018-03-14; First posted 2018-04-18 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Ischemic Heart Disease
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Intervention Model Description: In an online randomization module the randomization will be performed with permuted block randomization to 1:1 ratio.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No touch (Experimental): No touch technique. Patients are randomized to no touch vein harvesting. The technique is used as routine in Medical care by some hospitals.
  Interventions: Procedure: No touch technique
- Control (Other): Control technique. Patients are randomized to Control vein harvesting. The technique is used as routine in Medical care.
  Interventions: Procedure: Control technique

INTERVENTIONS:
Procedure: No touch technique — Veins for CABG is harvested with the no touch technique
  Arms: No touch
Procedure: Control technique — Veins for CABG is harvested with the Control technique.
  Arms: Control

SUMMARY:
The primary objective in this study is to investigate if vein grafts harvested and implanted with the non-touch technique are superior to conventional vein graft technique with respect to mid-term patency, in patients undergoing CABG surgery.

DETAILED DESCRIPTION:
Coronary artery bypass grafting (CABG) is the most common surgical procedure aimed against ischemic heart disease (IHD) in Sweden. Early and late success of CABG is the result of sustained patency of the bypass grafts. The choice of conduit (graft) for CABG has been shown to impact graft patency. The excellent early and late patency of in situ left internal thoracic artery (LITA) has stimulated the use of other arterial grafts, such as the radial artery (RA) and the right internal thoracic artery (RITA). However, target coronary vessels/lesions are limitations for the use of RITA and RA, and concerns regarding postoperative sternal wound infection with increases of early morbidity and mortality are reasons for limited use of bilateral ITA. The saphenous vein grafts (SVG), together with the left internal thoracic artery, are still the most commonly used conduits in CABG surgery.

Vein graft failure is associated with recurrence of angina and one of the primary reasons for reintervention, either by redo CABG or percutaneous coronary intervention (PCI). Early vein graft failure is not uncommon, and it was shown in the PREVENT IV multi-center trial6, that vein graft failure (occluded or stenosed) had occurred in 27% of all vein grafts at one year.

Despite this, SVG remains as an important conduit for most patients in contemporary bypass surgery and every effort should focus on promoting short and long-term patency of SVG. Previous studies by Souza have demonstrated that harvesting the SVG with a pedicle of surrounding tissue and without vein graft distension, the so-called "No touch" technique (NT), significantly improve patency compared with conventional technique i.e. stripping the vein of all adventitial tissue and distension prior to implantation. An international multi center randomized controlled clinical trial, (SUPERIOR SVG, NCT01047449) including 12 centers and 250 patients, was recently presented and showed favorable but not significant results for No touch vein grafts compared to conventional vein grafts. The protocol did not include cardiac computed tomography angiography (CCTA) for every patient which is an important difference compared to our planned study.

The major limitation regarding the putative benefit of NT technique of vein harvesting is that most of the data has all been derived from a single center. The surgical vein graft harvesting technique for NT grafts is more demanding. Therefore, there is a clear clinical equipoise to perform a multi-center randomized clinical trial to validate the excellent single-center results and determine whether the NT technique is reproducible, feasible and generalizable.

ELIGIBILITY:
Inclusion Criteria:

* first time CABG patients
* age up to 80 years at the time for inclusion
* need for at least one vein graft
* able to provide informed consent and accepted for isolated primary non-emergent CABG.

Exclusion Criteria:

* unable to use greater saphenous vein grafts (SVG) due to previous vein stripping or poor vein quality
* allergy to contrast dye
* renal failure with glomerular filtration rate (GFR)<15 ml/min
* coagulation disorders
* excessive risk of wound infection
* participation in other interventional trial on grafts
* any condition that seriously increases the risk of non-compliance or loss of follow-up

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 902 (Actual)
Dates: Start 2018-04-20 (Actual); Primary Completion 2023-09-19 (Actual); Study Completion 2023-11-17 (Actual)

PRIMARY OUTCOMES:
Saphenous vein grafts (SVGs) occluded/stenosed | Follow up period is from inclusion and surgery up to at least two years after.
  The proportion of patients with graft failure defined as: SVGs occluded/stenosed >50% on CCTA or has undergone percutaneous intervention to a vein graft or died within two years after CABG.

SECONDARY OUTCOMES:
Major adverse cardiac events (MACE) 1 | Follow up period is from inclusion and surgery up to at least two years after.
  The frequency of incidence of all cause death
MACE 2 | Follow up period is from inclusion and surgery up to at least two years after.
  The frequency of myocardial infarction
MACE 3 | Follow up period is from inclusion and surgery up to at least two years after.
  The frequency of repeated revascularization
Wound complications | Follow up period is from inclusion and surgery up to at least two years after.
  The frequency of incidence of postoperative leg wound complications from the harvesting site.
Vein-graft stenosis | Follow up period is from inclusion and surgery up to at least two years after.
  The frequency of non-significant vein graft stenosis (20-50%)
Perivascular inflammation | Follow-up period is from inclusion and surgery up to at least 2 years after.
  Perivascular fat attenuation index (FAIPVAT) around right coronary artery, no-touch saphenous vein grafts, and left internal mammary artery grafts

OTHER OUTCOMES:
Questions about wound healing | At 3 months and 2 years after CABG surgery.
  The questionnaires will be assessed by Telephone.
Questions about Quality of Life | At 2 years after CABG surgery.
  The patients will be interviewed about problems with angina (SAQ-7, Seattle Angina Questionnaire-7). The questionnaire will be assessed by telephone.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan James, Professor, Principal Investigator — Uppsala University Hospital
Locations (9):
- Aarhus, Aarhus, Denmark
- Sweden (8):
  - Göteborg, Gothenburg
  - Karlskrona, Karlskrona
  - Linköping, Linköping
  - Lund, Lund
  - Örebro, Sweden, Örebro
  - Karolinska Sjukhuset, Stockholm
  - Umeå, Umeå
  - Uppsala, Uppsala

REFERENCES:
- [Background] Loop FD, Lytle BW, Cosgrove DM, Stewart RW, Goormastic M, Williams GW, Golding LA, Gill CC, Taylor PC, Sheldon WC, et al. Influence of the internal-mammary-artery graft on 10-year survival and other cardiac events. N Engl J Med. 1986 Jan 2;314(1):1-6. doi: 10.1056/NEJM198601023140101. PMID 3484393
- [Background] Desai ND, Cohen EA, Naylor CD, Fremes SE; Radial Artery Patency Study Investigators. A randomized comparison of radial-artery and saphenous-vein coronary bypass grafts. N Engl J Med. 2004 Nov 25;351(22):2302-9. doi: 10.1056/NEJMoa040982. PMID 15564545
- [Background] Lytle BW, Blackstone EH, Loop FD, Houghtaling PL, Arnold JH, Akhrass R, McCarthy PM, Cosgrove DM. Two internal thoracic artery grafts are better than one. J Thorac Cardiovasc Surg. 1999 May;117(5):855-72. doi: 10.1016/S0022-5223(99)70365-X. PMID 10220677
- [Background] Parisian Mediastinitis Study Group. Risk factors for deep sternal wound infection after sternotomy: a prospective, multicenter study. J Thorac Cardiovasc Surg. 1996 Jun;111(6):1200-7. doi: 10.1016/s0022-5223(96)70222-2. PMID 8642821
- [Background] Guru V, Fremes SE, Tu JV. How many arterial grafts are enough? A population-based study of midterm outcomes. J Thorac Cardiovasc Surg. 2006 May;131(5):1021-8. doi: 10.1016/j.jtcvs.2005.09.036. Epub 2006 Apr 25. PMID 16678585
- [Background] Alexander JH, Hafley G, Harrington RA, Peterson ED, Ferguson TB Jr, Lorenz TJ, Goyal A, Gibson M, Mack MJ, Gennevois D, Califf RM, Kouchoukos NT; PREVENT IV Investigators. Efficacy and safety of edifoligide, an E2F transcription factor decoy, for prevention of vein graft failure following coronary artery bypass graft surgery: PREVENT IV: a randomized controlled trial. JAMA. 2005 Nov 16;294(19):2446-54. doi: 10.1001/jama.294.19.2446. PMID 16287955
- [Background] Souza DS, Dashwood MR, Tsui JC, Filbey D, Bodin L, Johansson B, Borowiec J. Improved patency in vein grafts harvested with surrounding tissue: results of a randomized study using three harvesting techniques. Ann Thorac Surg. 2002 Apr;73(4):1189-95. doi: 10.1016/s0003-4975(02)03425-2. PMID 11996262
- [Background] Souza DS, Johansson B, Bojo L, Karlsson R, Geijer H, Filbey D, Bodin L, Arbeus M, Dashwood MR. Harvesting the saphenous vein with surrounding tissue for CABG provides long-term graft patency comparable to the left internal thoracic artery: results of a randomized longitudinal trial. J Thorac Cardiovasc Surg. 2006 Aug;132(2):373-8. doi: 10.1016/j.jtcvs.2006.04.002. PMID 16872965
- [Background] Dashwood MR, Savage K, Dooley A, Shi-Wen X, Abraham DJ, Souza DS. Effect of vein graft harvesting on endothelial nitric oxide synthase and nitric oxide production. Ann Thorac Surg. 2005 Sep;80(3):939-44. doi: 10.1016/j.athoracsur.2005.03.042. PMID 16122459
- [Background] Dashwood MR, Savage K, Tsui JC, Dooley A, Shaw SG, Fernandez Alfonso MS, Bodin L, Souza DS. Retaining perivascular tissue of human saphenous vein grafts protects against surgical and distension-induced damage and preserves endothelial nitric oxide synthase and nitric oxide synthase activity. J Thorac Cardiovasc Surg. 2009 Aug;138(2):334-40. doi: 10.1016/j.jtcvs.2008.11.060. Epub 2009 Mar 10. PMID 19619776
- [Background] Samano N, Geijer H, Liden M, Fremes S, Bodin L, Souza D. The no-touch saphenous vein for coronary artery bypass grafting maintains a patency, after 16 years, comparable to the left internal thoracic artery: A randomized trial. J Thorac Cardiovasc Surg. 2015 Oct;150(4):880-8. doi: 10.1016/j.jtcvs.2015.07.027. Epub 2015 Jul 15. PMID 26282605
- [Result] Thelin S, Modrau IS, Duvernoy O, Dalen M, Dreifaldt M, Ericsson A, Friberg O, Holmgren A, Hostrup Nielsen P, Hultkvist H, Jensevik Eriksson K, Jeppsson A, Liden M, Nozohoor S, Ragnarsson S, Sartipy U, Ternstrom L, Themudo R, Vikholm P, James S. No-touch vein grafts in coronary artery bypass surgery: a registry-based randomized clinical trial. Eur Heart J. 2025 May 7;46(18):1720-1729. doi: 10.1093/eurheartj/ehaf018. PMID 39969129
- [Derived] Ragnarsson S, Janiec M, Modrau IS, Dreifaldt M, Ericsson A, Holmgren A, Hultkvist H, Jeppsson A, Sartipy U, Ternstrom L, Per Vikholm MD, de Souza D, James S, Thelin S. No-touch saphenous vein grafts in coronary artery surgery (SWEDEGRAFT): Rationale and design of a multicenter, prospective, registry-based randomized clinical trial. Am Heart J. 2020 Jun;224:17-24. doi: 10.1016/j.ahj.2020.03.009. Epub 2020 Mar 13. PMID 32272256